CLINICAL TRIAL: NCT00153972
Title: Dopamine Turnover Rate Measured With F-Dopa-PET as Surrogate Parameter for Diagnosis and Progression Analysis of Early Parkinson's Disease
Brief Title: Dopamine Turnover Rate as Surrogate Parameter for Diagnosis of Early Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Alexander Storch, Professor, Technische Universität Dresden
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 91052003
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2012-12-18 (Estimated); Status verified 2012-12

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Fluoro-Dopa-PET; Dopamine agonists; Cabergoline; Surrogate marker; Dopamine turnover
MeSH Terms: conditions — Parkinson Disease | interventions — Cabergoline; Levodopa

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Levodopa (Active Comparator): Levodopa 300 mg per day orally.
  Interventions: Drug: Cabergoline; Drug: Levodopa
- Cabergoline (Active Comparator): Cabergoline 3 mg per day orally.
  Interventions: Drug: Cabergoline; Drug: Levodopa

INTERVENTIONS:
Drug: Cabergoline
Drug: Levodopa

SUMMARY:
The study is designed to measure the difference of dopamine turnover rate measured by Fluoro-Dopa-PET in the putamen between patients with Parkinson's disease treated with cabergoline and levodopa for 3 months.

The study protocol includes an initial Fluoro-Dopa-PET scan before treatment and after three months double-blind treatment with cabergoline or levodopa.

The hypothesis for this study is that the dopamine turnover rate is a more sensitive marker for the early diagnosis of Parkinson's disease compared to the standard Fluoro-Dopa-PET measuring only the Fluoro-Dopa uptake into the striatum.

For the interventional part of the study, the hypothesis is that levodopa has larger effects on striatal dopamine turnover compared to dopamine agonists by providing more dopamine precursor. Enhancement of compensatory mechanisms for dopamine loss in early PD such as increased dopamine turnover could have several beneficial implications such as improvement or prolongation of symptomatic treatment responses, but might also produce therapeutic problems such as the development of levodopa-induced motor complications.

DETAILED DESCRIPTION:
The study is designed to measure the difference of dopamine turnover rate measured by Fluoro-Dopa-PET in the putamen between patients with Parkinson's disease treated with cabergoline and levodopa for 3 months.

The hypothesis for this study is that the dopamine turnover rate is a more sensitive marker for the early diagnosis of Parkinson's disease compared to the standard Fluoro-Dopa-PET measuring only the Fluoro-Dopa uptake into the striatum. The specific aim of the study was to estimate normal ranges and test-retest measures for various parameters characterising dopamine metabolism from a prolonged 18F-dopa positron emission tomography (PET) measurement using a reference tissue model and compare their value for the detection of early PD.

For the interventional part of the study, the hypothesis is that levodopa has larger effects on striatal dopamine turnover compared to dopamine agonists by providing more dopamine precursor. Enhancement of compensatory mechanisms for dopamine loss in early PD such as increased dopamine turnover could have several beneficial implications such as improvement or prolongation of symptomatic treatment responses, but might also produce therapeutic problems such as the development of levodopa-induced motor complications. The specific aim is to evaluate the effects of levodopa and the dopamine D2 agonist cabergoline on striatal dopamine turnover estimated as the inverse of the effective dopamine distribution volume ratio (EDVR) measured by 18F-dopa PET in de-novo PD.

The study protocol includes an initial Fluoro-Dopa-PET scan before treatment and after three months double-blind treatment with cabergoline or levodopa. This study is an investigator-blinded, randomized mono-center controlled phase IV study.

The main inclusion criteria are:

- Early (de novo) Parkinson's disease (Hoen & Yahr I and II), according to the UK brain bank criteria

The main exclusion criteria are:

* Current or past dopaminergic treatment
* Atypical parkinsonian syndromes
* Treatment with neuroleptics (present and past)

Methods:

* Fluoro-dopa-PET for measuring the dopamine turnover rate
* clinical investigations including parkinsonian rating scales (e.g. UPDRS, PDQ-39, etc.)
* olfactory tests

Study medication:

* Cabergoline (1 to 3 mg once per day)
* Levodopa/carbidopa (50 until 300 mg levodopa per day in one to three dosages)

ELIGIBILITY:
Inclusion Criteria:

* Early (de novo) Parkinson's disease (Hoen & Yahr I and II), according to the UK brain bank criteria

Exclusion Criteria:

* Current or past dopaminergic treatment
* Atypical parkinsonian syndromes
* Treatment with neuroleptics (present and past)
* Pregnancy

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-02; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Difference of dopamine turnover rate measured by Fluoro-Dopa-PET in the putamen between patients with Parkinson's disease treated with cabergoline and levodopa for 3 months.

SECONDARY OUTCOMES:
Changes of clinical outcome measured with parkinsonian rating scales (UPDRS, PDQ-39, ESS, olfactory function)

CONTACTS AND LOCATIONS:
Overall Officials: Heinz Reichmann, MD, Principal Investigator — Technical University of Dresden
Locations (2):
- Germany (2):
  - Department of Neurology at the Technical University of Dresden, Dresden, Saxony
  - Department of Nuclear Medicine at the Technical University of Dresden, Dresden, Saxony

REFERENCES:
- [Result] Oehme L, Perick M, Beuthien-Baumann B, Wolz M, Storch A, Lohle M, Herting B, Langner J, van den Hoff J, Reichmann H, Kotzerke J. Comparison of dopamine turnover, dopamine influx constant and activity ratio of striatum and occipital brain with (1)(8)F-dopa brain PET in normal controls and patients with Parkinson's disease. Eur J Nucl Med Mol Imaging. 2011 Aug;38(8):1550-9. doi: 10.1007/s00259-011-1819-8. Epub 2011 May 7. PMID 21553090
- See also: Homepage of principle location — http://www.neuro.med.tu-dresden.de